CLINICAL TRIAL: NCT03625570
Title: Power Training Combined With Interval Treadmill Training to Improve Walking Activity in Cerebral Palsy (PT³)
Brief Title: Power Training Combined With Interval Treadmill Training
Acronym: PT³
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD091089 (NIH); R01HD091089 (NIH)
Record Dates: First submitted 2018-08-01; First posted 2018-08-10 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy; Central Nervous System Diseases; Brain Damage, Chronic
Keywords: muscle weakness; muscle power; resistance training; treadmill training
MeSH Terms: conditions — Cerebral Palsy; Central Nervous System Diseases; Brain Damage, Chronic; Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT³ (Experimental): Power Training combined with interval treadmill training
  Interventions: Behavioral: Power training combined with interval treadmill training
- Traditional training (Active Comparator): Strength training combined with traditional treadmill training
  Interventions: Behavioral: Strength training combined with traditional treadmill training

INTERVENTIONS:
Behavioral: Power training combined with interval treadmill training — Training will consist of unilateral and bilateral leg presses, targeting the quadriceps, hip extensors, and plantarflexors according to resistance training guidelines for muscle power training. The interval treadmill training portion will include short-bursts (30 seconds) of high speed walking intervals alternating with 30 seconds of low to moderate speed walking for a total of 30 minutes. Participants will train 3 x per week for 8 weeks. Total duration of each session will be approximately 1 hour.
  Arms: PT³
Behavioral: Strength training combined with traditional treadmill training — Training will consist of unilateral and bilateral leg presses, targeting the quadriceps, hip extensors, and plantarflexors following the dosing and resistance training guidelines for muscle strength. Traditional treadmill training will consist of walking at steady-state speeds for 30 minutes. Participants will train 3 x per week for 8 weeks. Total duration of each session will be approximately 1 hour.
  Arms: Traditional training

SUMMARY:
Ambulatory children with cerebral palsy (CP) experience walking limitations which negatively influence their ability to physically participate in day to day life. The investigators propose that impaired muscle power generation is the key limiting factor affecting walking activity and participation. This proposal represents a combined approach where participants undergo resistance training for muscle power generation in combination with locomotor treadmill training that is based on typical pediatric walking and activity patterns rather than adult protocols, which are endurance or time-based. Therefore, the primary objective of this randomized controlled trial is to determine the effect of lower extremity Power Training combined with interval Treadmill Training (PT³) on functional walking capacity and community-based activity and participation in children with CP. We hypothesize that remediating the most pronounced muscle performance impairment (i.e., muscle power) with power training combined with a task- specific approach to walking that is developmentally appropriate will have a significant effect on walking capacity and performance.

DETAILED DESCRIPTION:
The primary purpose of this randomized controlled trial is to test the effect of Power Training combined with interval Treadmill Training (PT³) on walking capacity and performance in children with CP with walking limitations. To identify key muscular mechanisms associated with improved walking mobility, the effects of PT³ on muscle performance and architecture will be examined. The premise of the PT³ protocol is that a combined impairment and task-specific approach that is developmentally appropriate and targets muscle power deficits specifically, is necessary to drive changes in both clinic and community-based walking activity.

In this randomized multi-site clinical trial, 48 ambulatory participants with CP will receive either PT³ or an equivalent dosage of traditional strength training combined with traditional treadmill training (comparison group) for 24 sessions, 3 times per week for 8 weeks. Outcomes will be collected at baseline and immediately post-treatment. Short and long-term retention effects will be assessed at 2 and 6 months post.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral spastic Cerebral Palsy (CP)
* Age 10 to 17 years inclusive
* GMFCS levels I, II, or III

Exclusion Criteria:

* Orthopedic or neurosurgery less than 12 months prior to enrollment
* Injection therapies (phenol, botulinum toxin) less than 3 months prior to enrollment
* Lacking greater than 25 degrees of knee extension

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle G Moreau, PT, PhD, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (2):
- United States (2):
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at two sites (academic medical center and a children's hospital). Participants were recruited from the surrounding community and regional tertiary pediatric care centers.
Pre-assignment Details: Of the 44 enrolled participants, 43 were randomized. 1 participant was excluded prior to randomization due to the inability to cooperate and complete baseline assessments.
Groups:
- PT³ (Power Training Combined With Interval Treadmill Training): Power Training combined with interval treadmill training
  Power training combined with interval treadmill training: Training will consist of unilateral and bilateral leg presses, targeting the quadriceps, hip extensors, and plantarflexors according to resistance training guidelines for muscle power training. The interval treadmill training portion will include short-bursts (30 seconds) of high speed walking intervals alternating with 30 seconds of low to moderate speed walking for a total of 30 minutes. Participants will train 3 x per week for 8 weeks. Total duration of each session will be approximately 1 hour.
- Traditional Training (Strength Training Combined With Traditional Treadmill Training): Strength training combined with traditional treadmill training
  Strength training combined with traditional treadmill training: Training will consist of unilateral and bilateral leg presses, targeting the quadriceps, hip extensors, and plantarflexors following the dosing and resistance training guidelines for muscle strength. Traditional treadmill training will consist of walking at steady-state speeds for 30 minutes. Participants will train 3 x per week for 8 weeks. Total duration of each session will be approximately 1 hour.
Period: Primary Endpoint - Immediate Post
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Traditional Treadmill Training)
Started | 23 | 20
Completed (Completed Intervention) | 20 | 18
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — PI decision; unable to perform exercises | 1 | 0
Not completed — Withdrawn; COVID-19 shut down | 0 | 1
Period: Secondary Endpoint - 2 Months Post
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Traditional Treadmill Training)
Started | 20 | 18
Completed (2mo. Post Follow-up) | 18 | 17
Not Completed | 2 | 1
Period: Secondary Endpoint - 6 Months Post
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Traditional Treadmill Training)
Started | 18 | 17
Completed | 18 | 16
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Traditional Training (Strength Training Combined With Treadmill Training): Strength training combined with traditional treadmill training
  Strength training combined with traditional treadmill training: Training will consist of unilateral and bilateral leg presses, targeting the quadriceps, hip extensors, and plantarflexors following the dosing and resistance training guidelines for muscle strength. Traditional treadmill training will consist of walking at steady-state speeds for 30 minutes. Participants will train 3 x per week for 8 weeks. Total duration of each session will be approximately 1 hour.
- Total: Total of all reporting groups
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training) | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.07 (2.18) | 13.77 (2.55) | 13.39 (2.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 13 | 15 | 28
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 23 | 20 | 43
GMFCS Level [Count of Participants; unit: Participants] — Gross Motor Function Classification System (GMFCS) Level. Levels range from I to III for this study; however, the entire scale ranges from I to V. GMFCS levels are ordinal with lower levels indicating higher functioning or gross motor function ability, i.e, level I represents the highest level of function and level V represents the lowest level of function.
  Participants
    GMFCS Level I | 5 | 7 | 12
    GMFCS Level II | 14 | 12 | 26
    GMFCS Level III | 4 | 1 | 5
Body mass [Mean (Standard Deviation); unit: kilograms (kg)] | 44.43 (12.22) | 48.40 (19.86) | 46.28 (16.15)
Height [Mean (Standard Deviation); unit: meters] | 1.50 (0.12) | 1.53 (0.15) | 1.516 (0.14)
Enrollment Site [Count of Participants; unit: Participants] — LSUHSC - Louisiana State University Health Sciences Center, New Orleans, LA, USA SCRI - Seattle Children's Research Institute, Seattle, WA, USA
  Participants
    LSUHSC | 11 | 10 | 21
    SCRI | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-selected Gait Speed (Normalized)
Description: Calculated from the 10 meter walk test in meters/second at self-selected speed and then normalized by stature to yield non-dimensional units. Higher values represent faster gait speeds.
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: The a priori analytic approach included all participants in the primary analysis with the first (baseline) and second assessments.
  Least squares (LS) means adjusted for baseline and 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
dimensionless | -0.0010 (0.0096) | 0.0163 (0.0100)

2. Primary Outcome: Change in Fast Gait Speed (Normalized)
Description: Calculated from the 10 meter walk test in meters/second at fast walking speed and then normalized by stature to yield non-dimensional units. Higher values equal faster gait speeds.
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: The a priori analytic approach included all participants in the primary analysis with the first (baseline) and second assessments.
  LS Means adjusted for baseline and 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
dimensionless | 0.0204 (0.0074) | 0.0093 (0.0080)

3. Primary Outcome: Change in Peak Power
Description: Lower extremity peak power produced during a power leg press test averaged over 5 trials; product of force x velocity; adjusted for sled angle and body mass
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: The a priori analytic approach included all participants in the primary analysis with the first (baseline) and second assessments.
  LS Means adjusted for 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: watts
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
watts | 71.21 (18.71) | 19.19 (19.83)

4. Primary Outcome: Change in Average Strides Per Day
Description: Average number of strides walked per day captured by Step Watch accelerometer as worn for a minimum of 4 days
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: strides/day
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
strides/day | -95.84 (284.85) | -16.03 (318.79)

5. Secondary Outcome: Change in Self-selected Gait Speed (Normalized)
Description: Calculated from the 10 meter walk test in meters/second at self-selected speed and then normalized by stature to yield non-dimensional units. Higher values equal faster speeds.
Time Frame: Baseline and 2 months post training (16 weeks post baseline)
Population: LS Means adjusted for baseline and 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 18 | 17
dimensionless | 0.0156 (0.0092) | 0.0144 (0.0092)

6. Secondary Outcome: Change in Fast Gait Speed (Normalized)
Description: Calculated from the 10 meter walk test in meters/second at fast walking speed and then normalized by stature to yield non-dimensional units. Higher values equal faster speeds.
Time Frame: Baseline and 2 months post training (16 weeks post baseline)
Population: LS Means adjusted for baseline and 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: dimensionless
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 18 | 17
dimensionless | 0.0528 (0.0125) | 0.0226 (0.0127)

7. Secondary Outcome: Change in Peak Power
Description: as for outcome 3
Time Frame: Baseline and 2 months post training (16 weeks post baseline)
Population: LS Means adjusted for 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: watts
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 18 | 16
watts | 57.9248 (22.3544) | 1.5342 (23.4939)

8. Secondary Outcome: Change in Average Strides Per Day
Description: Average number of strides walked per day captured by Step Watch accelerometer as worn for a minimum of 4 days
Time Frame: Baseline and 2 months post training (16 weeks post baseline)
Population: LS Means adjusted for 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: strides/day
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 18 | 13
strides/day | -139.77 (324.13) | -299.82 (373.20)

9. Secondary Outcome: Change in One Minute Walk Test
Description: Distance covered while walking as fast as possible for 1 minute measured in meters
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: LS Means adjusted for baseline and 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
meters | 8.349 (2.637) | 7.750 (2.764)

10. Secondary Outcome: Change in Cross-sectional Area
Description: Cross-sectional area of rectus femoris taken at 50% distance between anterior superior iliac spine and apex of patella using 2D Bmode Ultrasound imaging in cm^2; Average of Right and Left Sides
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: LS Means adjusted for 3 covariates (Age group; Site; GMFCS level) and side tested (left and right)
Measure: Least Squares Mean (Standard Error); unit: cm^2
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 17 | 18
cm^2 | 0.3390 (0.0667) | 0.2692 (0.0684)

11. Secondary Outcome: Change in Isokinetic Muscle Strength of Knee Extensors
Description: Isokinetic dynamometer (Biodex System 3/4) according to published standard procedures for isokinetic strength. Calculated for knee extensors at 60 degrees/second in newton-meters
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: LS means adjusted for 3 covariates (Age group; Site; GMFCS level) and side tested (left and right)
Measure: Least Squares Mean (Standard Error); unit: Nm
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
Nm | 3.8778 (3.0255) | 2.1524 (3.1937)

12. Secondary Outcome: Change in Walking Intensity at Medium and High Stride Rates (Strides/Minute)
Description: Average strides/day at medium (31 to 60 stride/min) and high (> 60 stride/min) stride rates as captured by Step Watch accelerometer as worn for a minimum of 4 days
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: LS Means adjusted for 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: strides/minute
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 19 | 16
strides/minute | 0.01313 (0.0289) | -0.06635 (0.0323)

13. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System Physical Function-Mobility (PROMIS v2.0 Pediatric Profile 49 - Physical Function-Mobility)
Description: Patient-Reported Outcomes Measurement Information System (PROMIS); The PROMIS item bank was developed from patient-reported outcome measures that indicate patients' state of well-being and functional abilities. The results of the Physical Function-Mobility domain are reported here as the Change in the T-score from baseline to 8-10wks post baseline. The T-score is a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean. A higher PROMIS T-score represents more of the concept being measured so for a positive concept, such as Physical Function-Mobility, a higher T-score or 'change' in the T-score represents higher physical functioning and mobility.
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: Least squares (LS) means adjusted for 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
T-score | 2.229 (1.72) | 2.792 (1.83)

14. Secondary Outcome: Change in 1RM (Muscle Strength)
Description: 1repetition maximum (1RM) testing on a leg press reported in lbs; external load reported after adjusting for the angle of the press
Time Frame: Baseline and immediate post training (8-10 weeks post baseline)
Population: LS Means adjusted for baseline and 3 covariates (Age group; Site; GMFCS level)
Measure: Least Squares Mean (Standard Error); unit: lbs
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
Number analyzed (Participants) | 20 | 18
lbs | 54.568 (13.031) | 49.961 (14.263)

ADVERSE EVENTS:
Time Frame: From enrollment to 6 months post-intervention (32 weeks post baseline)
Arm/Group | PT³ (Power Training Combined With Interval Treadmill Training) | Traditional Training (Strength Training Combined With Treadmill Training)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/20
Other Adverse Events (participants affected / at risk) | 7/23 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PT³ (Power Training Combined With Interval Treadmill Training) (N=23) | Traditional Training (Strength Training Combined With Treadmill Training) (N=20)
Ventriculoperitoneal (VP) shunt revision (Not Related to the Study) (Surgical and medical procedures) | 1 (1) | 0 (0) — Ventriculoperitoneal (VP) shunt revision was needed that was determined to be "Not Related to the Study"
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PT³ (Power Training Combined With Interval Treadmill Training) (N=23) | Traditional Training (Strength Training Combined With Treadmill Training) (N=20)
blisters (Skin and subcutaneous tissue disorders) | 2 | 3 — blisters on either hands or feet
dizziness (Ear and labyrinth disorders) | 1 | 0
exercise-induced asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
knee or leg pain (General disorders) | 1 | 4
muscle soreness (General disorders) | 1 | 1
muscle spasm (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03625570/Prot_SAP_000.pdf